CLINICAL TRIAL: NCT06440772
Title: Assessing Fluid Intolerance Using Portal Vein Pulsatility Index Post-Passive Leg Raising Test in Fluid Responders: A Prospective Cohort Study
Brief Title: Portal Vein Pulsatility Index to Assess Fluid Intolerance
Status: Completed | Type: Observational
Sponsor: Institutul de Urgenţă pentru Boli Cardiovasculare Prof.Dr. C.C. Iliescu (Other)
Responsible Party: Principal Investigator, Balan Ion Cosmin, Principal Investigator, Institutul de Urgenţă pentru Boli Cardiovasculare Prof.Dr. C.C. Iliescu
Other Study IDs: 6066/21.02.2023
Record Dates: First submitted 2024-05-30; First posted 2024-06-04 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Venous Congestion
Keywords: congestion; portal vein pulsatility; ultrasound; fluid responsiveness; fluid tolerance
MeSH Terms: conditions — Hyperemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tolerant Fluid Responders: Patients who are both responsive and tolerant to fluid.
  Interventions: Drug: Ringer's Lactate Crystalloid Solutions

INTERVENTIONS:
Drug: Ringer's Lactate Crystalloid Solutions — 7 ml/kg ml of Ringer's Lactate is given in 10 min amongst initially tolerant fluid responders.
  Other Names: Fluid challenge

SUMMARY:
This study uses the portal vein pulsatility index (PVPI) to assess fluid intolerance amongst fluid responders.

DETAILED DESCRIPTION:
This prospective observational study aims to use the portal vein pulsatility index (PVPI) to assess fluid intolerance in fluid responders. The investigators will enroll mechanically ventilated postoperative adult patients within 6 hours of ICU admission after cardiac surgery. Patients will undergo a Passive Leg Raising (PLR) test and Left Ventricular Outflow Tract (LVOT) recording using transthoracic echocardiography. The main objective is to predict fluid intolerance after a fluid challenge of 7 ml/kg Ringer Lactate over 10 minutes in initially tolerant fluid responders.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent.
* Mechanically ventilated patients within 6 hours after ICU admission following surgery who are considered for fluid administration to optimize haemodynamics.
* Sinus rhythm.

Exclusion Criteria:

* A condition known to interfere with portal vein flow assessment or interpretation (liver cirrhosis or chronic hepatic disease, suprahepatic or portal vein thrombosis).
* Any mechanical circulatory support.
* Cardiac transplant.
* Poor transthoracic echocardiographic window.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated postoperative adult patients after cardiac surgery within 6 hours after intensive care unit admission.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Fluid Intolerance | 10 minutes after 7 ml/kg Ringer's Lactate
  A portal vein pulsatility index greater than 50%, calculated as (Vmax - Vmin) / Vmax, with no upper limit and 0% as the minimum limit. Higher values indicate worse outcomes. Ultrasonographic portal spectral waveform was used to measure Vmax and Vmin.

CONTACTS AND LOCATIONS:
Overall Officials: Cosmin Balan, PhD, Principal Investigator — "Prof CC Iliescu" Emergency Institue for Cardiovascular Diseases; Serban-Ion Bubenek-Turconi, Professor, Study Chair — "Prof CC Iliescu" Emergency Institue for Cardiovascular Diseases
Locations (1):
- "Prof CC Iliescu" Emergency Institue for Cardiovascular Diseases, Bucharest, Romania

REFERENCES:
- [Derived] Balan C, Morosanu B, Fodoroiu A, Dobre V, Dumitrache A, Barbulescu RT, Valeanu L, Robu C, Boros C, Nica A, Wong A, Corradi F, Grintescu IM, Bubenek-Turconi SI. Decoding portal vein pulsatility: hemodynamic determinants in a post-hoc analysis of a prospective observational trial. Ann Intensive Care. 2025 Jun 14;15(1):81. doi: 10.1186/s13613-025-01498-0. PMID 40515791
- [Derived] Morosanu B, Balan C, Boros C, Dazzi F, Wong A, Corradi F, Bubenek-Turconi SI. Incidence, predictability, and outcomes of systemic venous congestion following a fluid challenge in initially fluid-tolerant preload-responders after cardiac surgery: a pilot trial. Crit Care. 2024 Oct 22;28(1):339. doi: 10.1186/s13054-024-05124-6. PMID 39439007